CLINICAL TRIAL: NCT03271671
Title: A Randomized Controlled Trial Comparing Non-invasive Ventilation (NIV) With Pressure Support Ventilation (PSV) Versus Neurally Adjusted Ventilator Assist (NAVA) During Acute Respiratory Failure (ARF)
Brief Title: Pressure Support Ventilation (PSV) Versus Neurally Adjusted Ventilator Assist (NAVA) During Acute Respiratory Failure (ARF)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Inderpaul singh, Assistant Professor, Department of Pulmonary Medicine, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TRB2447/1/7/17
Record Dates: First submitted 2017-09-01; First posted 2017-09-05 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Respiratory Failure
Keywords: neurally adjusted ventilator assist; Pressure support ventilation; non invasive ventilation; niv
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial comparing two modes of non invasive ventilation
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PSV (Active Comparator): Pressure support ventilation
  Interventions: Other: PSV during Non invasive ventilation
- NAVA (Experimental): Neurally adjusted ventilator assist
  Interventions: Other: NAVA during Non invasive ventilation

INTERVENTIONS:
Other: NAVA during Non invasive ventilation — NIV during respiratory failure
  Arms: NAVA
Other: PSV during Non invasive ventilation — PSV during respiratory failure
  Arms: PSV

SUMMARY:
Acute respiratory failure (ARF) is a life-threatening emergency which occurs due to impaired gas exchange. In the US, the number of hospitalisations owing to acute respiratory failure was 1,917,910 in the year 2009.(1) The incidence of ARF requiring hospitalization was 137.1 per 100,000 population.(2) In ARF due to chronic obstructive pulmonary disease (COPD) and cardiogenic pulmonary edema, non-invasive ventilation (NIV) has been shown to be beneficial. NIV also has several advantages over invasive mechanical ventilation. These include, avoidance of endotracheal intubation and its attendant complications like airway injury, nosocomial infections, and possibly shorter duration of intensive care unit (ICU) stay.(3, 4) The success of NIV depends on several factors like the etiology of the respiratory failure, careful monitoring by the treating physician, and also adequate cooperation of patient. Better synchrony of the patient's spontaneous breaths with the ventilator-delivered breaths may lead to better patient cooperation and thereby, better clinical outcomes. Patient-ventilator asynchrony (PVA) leads to dyspnea, increased work of breathing, and prolonged duration of mechanical ventilation.(5) Pressure support ventilation (PSV) is one of the commonest mode used during NIV. In a prospective multicenter observational study, severe asynchrony (defined as an asynchrony index of >10 %) was seen in 43% of patients of patients with ARF ventilated by NIV with the conventional PSV mode.(6) Neurally adjusted ventilator assist (NAVA) is new mode of ventilation which utilizes the electrical activity of the diaphragm to deliver the breath.(7) During NAVA, breath is delivered when the patient's diaphragm starts contracting. Further, the amount of pressure support given during the breath is proportional to the strength of the electrical signal from the diaphragm. Finally, NAVA also terminates the breath when the electrical activity of the diaphragm wanes. NAVA has been shown to avoid over-assistance, decrease intrinsic positive end-expiratory pressure (PEEP), and minimize wasted efforts.(8) Hence, NAVA may play a major role in improving patient-ventilator synchrony.

In a pooled analysis of studies comparing NAVA with PSV during NIV, it was shown that the use of NAVA significantly improved patient-ventilator synchrony.(9) However, so far, no clinical trial has demonstrated that this improvement in synchrony translates into better clinical outcomes. In this randomized controlled clinical trial, we intend to compare the rates of NIV failure and mortality between NAVA and PSV in subjects with acute respiratory failure managed with NIV.

DETAILED DESCRIPTION:
NIV is mode of ventilation wherein positive pressure ventilation is delivered by non-invasive interface like nasal mask, face mask, nasal plugs or helmet avoiding invasive interface by endotracheal intubation or by tracheostomy. In 1980s NIV by mask was used with success in patients of obstructive sleep apnea and later on in neuromuscular respiratory failure. Use of NIV has increased subsequently over next 20 years with overall first line NIV being used upto 23% (10) NIV is definitely useful as first line of management in COPD exacerbation, cardiogenic pulmonary edema, post extubation respiratory failure and is also worth trial with conflicting data in cases of acute hypoxemic respiratory failure due to pneumonia, ARDS.

In cases of acute exacerbation of COPD, NIV improves clinical outcomes.(11-13) In a metaanalysis by Ram FS et al which included 14 RCT and 758 patients which showed decreased mortality(11 vs 21%), intubation rate(16 vs 33%) and treatment failure(20 vs 42%)(12). Similarly, there is high quality evidence supporting use in cardiogenic pulmonary edema showing to improve respiratory parameters and decrease intubation rates (14-17). A meta-analysis of 32 studies including 2916 patients in 2013 by Vital FM et al showed that NIV reduces in hospital mortality compared to standard medical care(RR 0.66, 95% CI 0.48 - 0.89)(14) NAVA as mode of ventilation was developed after initial landmark study "neural control of mechanical ventilation in respiratory failure" was published in 1998 by Sinderby(7). It was later on introduced on the servo-i ventilator in 2007. NAVA is a kind of pressure assist ventilation using electrical activity of diaphragm and thus the neural output to initiate the breath, regulate the assist level and cycle off the breath.

In study by Piquilloud et al of 13 patients which compared NAVA with PSV during NIV there was significant difference in asynchronies. Trigger delay (Td) was reduced with NAVA to 35 ms (IQR 31-53 ms) versus 181 ms (122 - 208 ms). Also, there were no premature or delayed cycling, ineffective efforts in the NAVA group. Asynchrony index (AI) with NAVA was 4.9% (2.2 - 10.5%) compared to 15.8% (5.5 - 49.6%) with PSV (20)In a recent meta-analysis comparing PSV with NAVA during NIV by Inderpaul et al which included 9 studies with 96 subjects including both adult and paediatric patients showed that asynchronies were more in PSV than in NAVA in both adult and paediatric studies. The overall pooled mean difference of asynchrony index was 28.02(95% CI, 11.61 - 44.42). also the risk of severe asynchrony was 3.4 % times higher in PSV compared to NAVA group.(9) NAVA mode of ventilation in previous studies has shown to decrease asynchrony with ventilator, mainly reducing ineffective efforts, cycling delays. Ineffective efforts may occur due to presence of intrinsic PEEP which in turn is more common during prolonged insufflations and at high levels of assist. Ineffective efforts may also occur with weak inspiratory efforts which may occur during states of high respiratory drive. NAVA uses electrical activity of diaphragm to trigger a breath and there is marked difference in improving synchrony with studies reporting no wasted efforts when compared to PSV mode. In a study by Vignaux et al showed that during conventional NIV, 40 % of the patients experience asynchrony and the rate of asynchrony correlated with leakage(6). In NAVA mode of ventilation assistance is delivered based upon the neural trigger and hence is not affected by leaks.

In a pooled analysis of studies comparing NAVA with PSV during NIV, it was shown that the use of NAVA significantly improved patient-ventilator synchrony.(9) However, so far, no clinical trial has demonstrated that this improvement in synchrony translates into better clinical outcomes. In this randomized controlled clinical trial, we intend to compare the rates of NIV failure and mortality between NAVA and PSV in subjects with acute respiratory failure managed with NIV.

ELIGIBILITY:
Inclusion Criteria:

1. Respiratory rate >30 per minute
2. Arterial blood gas analysis showing a PaCO2 >45 mmHg and pH <7.35
3. PaO2/FiO2 ratio < 300
4. Use of accessory muscles of respiration or paradoxical respiration

Exclusion Criteria:

1. Age <18 years or >75 years
2. Pregnancy
3. PaO2/FiO2 ratio ≤100
4. Hypotension (systolic blood pressure <90 mmHg)
5. Severe impairment of consciousness (Glasgow coma scale score <8)
6. Inability to clear respiratory secretions (Airway care score [ACS] ≥12)(27)
7. Abnormalities that preclude proper fit of the NIV interface (agitated or uncooperative patient, facial trauma or burns, facial surgery, or facial anatomical abnormality)
8. Subjects who have an artificial airway like tracheostomy tube or T-tube
9. Contraindications for insertion of naso-/orogastric feeding tube (facial/nasal trauma, recent upper airway surgery, esophageal surgery, esophageal varices, upper gastrointestinal bleeding)
10. More than two organ failures
11. Unwillingness to undergo placement of nasogastric catheter
12. Known phrenic nerve lesions
13. Suspected diaphragmatic weakness
14. Patient already on home NIV therapy for chronic respiratory failure
15. Application of NIV for more than one hour for the current illness
16. Failure to provide informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Rates of NIV failures | 28 days
  NIV will be deemed to have failed if the patient gets intubated or is reinitiated on NIV within 48 hours of discontinuation of NIV
28-day mortality | 28 days
  28-day mortality including ICU and hospital deaths will be assessed

SECONDARY OUTCOMES:
Time to successful weaning | 28 days
  Time to successful weaning will be defined as the duration between initiation of NIV and successful weaning from NIV.
Time to NIV failure | 28 days
  Time to NIV failure will be calculated as the duration between initiation of NIV and the event which lead to NIV failure.
Total duration of mechanical ventilation (both non-invasive and invasive) | 28 days
  Total duration of mechanical ventilation will be calculated as the total duration spent on NIV and IMV by the patient.
Length of ICU and hospital stay | 28 days
  The length of ICU and hospital stay of the patient will also be assessed.
Patient's level of comfort during NIV using VAS | 28 days
  The patient's level of comfort while undergoing NIV will be assessed using a similar VAS. These assessments will be made every day till day 5 or till the patient is weaned off NIV, whichever is earlier.
Physician's level of comfort while using the assigned NIV strategy using VAS | 28 days
  The physician's level of comfort while using the two different modes of NIV will be assessed using a visual analogue scale (VAS). The assessment will be obtained from the treating physician at each shift.

CONTACTS AND LOCATIONS:
Overall Officials: Inderpaul S Sehgal, MD,DM, Principal Investigator — PGIMER,Chandigarh
Locations (1):
- Respiratory ICU, Post Graduate Institue of Medical Education and Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Undecided
Complete protocol and individual patient data after publication of results

REFERENCES:
- [Background] Stefan MS, Shieh MS, Pekow PS, Rothberg MB, Steingrub JS, Lagu T, Lindenauer PK. Epidemiology and outcomes of acute respiratory failure in the United States, 2001 to 2009: a national survey. J Hosp Med. 2013 Feb;8(2):76-82. doi: 10.1002/jhm.2004. Epub 2013 Jan 18. PMID 23335231
- [Background] Behrendt CE. Acute respiratory failure in the United States: incidence and 31-day survival. Chest. 2000 Oct;118(4):1100-5. doi: 10.1378/chest.118.4.1100. PMID 11035684
- [Background] Peter JV, Moran JL, Phillips-Hughes J, Warn D. Noninvasive ventilation in acute respiratory failure--a meta-analysis update. Crit Care Med. 2002 Mar;30(3):555-62. doi: 10.1097/00003246-200203000-00010. PMID 11990914
- [Background] Girou E, Schortgen F, Delclaux C, Brun-Buisson C, Blot F, Lefort Y, Lemaire F, Brochard L. Association of noninvasive ventilation with nosocomial infections and survival in critically ill patients. JAMA. 2000 Nov 8;284(18):2361-7. doi: 10.1001/jama.284.18.2361. PMID 11066187
- [Background] Georgopoulos D, Prinianakis G, Kondili E. Bedside waveforms interpretation as a tool to identify patient-ventilator asynchronies. Intensive Care Med. 2006 Jan;32(1):34-47. doi: 10.1007/s00134-005-2828-5. Epub 2005 Nov 9. PMID 16283171
- [Background] Vignaux L, Vargas F, Roeseler J, Tassaux D, Thille AW, Kossowsky MP, Brochard L, Jolliet P. Patient-ventilator asynchrony during non-invasive ventilation for acute respiratory failure: a multicenter study. Intensive Care Med. 2009 May;35(5):840-6. doi: 10.1007/s00134-009-1416-5. Epub 2009 Jan 29. PMID 19183949
- [Derived] Prasad KT, Gandra RR, Dhooria S, Muthu V, Aggarwal AN, Agarwal R, Sehgal IS. Comparing Noninvasive Ventilation Delivered Using Neurally-Adjusted Ventilatory Assist or Pressure Support in Acute Respiratory Failure. Respir Care. 2021 Feb;66(2):213-220. doi: 10.4187/respcare.07952. Epub 2020 Sep 1. PMID 32873750